CLINICAL TRIAL: NCT05012150
Title: A Pilot Study in Endoscopic Therapy on Quality of Life and Pain in Chronic Pancreatitis: The EQuiPP Study
Brief Title: A Pilot Study in Endoscopic Therapy on Quality of Life and Pain in Chronic Pancreatitis
Acronym: EQuiPP
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Mitchell Ramsey, Assistant Professor, Ohio State University
Other Study IDs: 2020H0410
Record Dates: First submitted 2021-07-27; First posted 2021-08-19 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pancreatitis
Keywords: ERCP; ESWL; quality of life; quantitative sensory testing; celiac plexus block; pancreatic duct stricture; pancreatic duct stenting; pancreatic fluid collection
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Stool, Saliva, and Pancreatic Fluid (juice) will be collected before and after endotherapy and stored in our Biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a prospective study designed to assess the effect of pancreatic endotherapy on quality of life, pain levels, pancreatic exocrine function, and endocrine function.

DETAILED DESCRIPTION:
Pancreatic endotherapy represents a potential treatment modality for patients with painful chronic pancreatitis. While pancreatic endotherapy is commonly performed, the effect of chronic pancreatitis on patient-centered outcomes remains poorly studied. Furthermore, the effect of endotherapy on pancreatic endocrine and exocrine are largely unknown. This study therefore aims to prospective observe patients with chronic pancreatitis after endotherapy is performed to better understand how it affects patient-centered outcomes such as pain and quality of life and pancreatic function. In doing so, the study also hopes to be able to predict which patients with chronic pancreatitis will benefit from pancreatic endotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pancreatitis (as defined by the American Pancreatic Association Guidelines)
* Presence of Pain
* Referred for pancreatic endotherapy

Exclusion Criteria:

* Prior pancreatic endotherapy
* Prior pancreatic surgery
* Pregnant females
* Subjects unable to consent
* Imprisoned individuals

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with painful chronic pancreatitis who are being referred for pancreatic endotherapy will be eligible for participation in this study. Subjects who have already had prior endotherapy or surgery, however, will be excluded.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Pancreatitis-Specific Quality of Life | 12 months post-completion of endotherapy
  Quality of life will be primarily assessed using the PANcreatitis Quality of Life Instrument (PANQOLI). Quality of life will be assessed before and after endotherapy (1, 3, 6, and 12 months). This instrument is based on a 0-87 scale with higher scores representing improved quality of life.
Feasibility of Micro-Longitudinal Daily Pain Assessment | 30-day post-procedure period
  Pain will be assessed using daily pain diaries with the Brief Pain Inventory (BPI). These will be utilized to create short-term pain trajectories for subjects at baseline and post-procedure. This pain inventory includes 9 pain items graded on 0-10 scale with 10 being the worst pain.

SECONDARY OUTCOMES:
Overall Quality of Life | 12 months post-completion of endotherapy
  Quality of life will be primarily assessed using the PROMIS-29 instrument. Quality of life will be assessed before and after endotherapy (1, 3, 6, and 12 months). The PROMIS-29 instrument incorporates 7 domains: physical functioning, fatigue, pain interference, depression, anxiety, ability to participate in social roles and activities, and sleep disturbance. Each of these domains have a score 0-40 with higher scores representing worse quality of life in these domains. There are also 2 summary scores: Physical Health and Mental Health. Z-scores are calculated for these two summary scores with lower scores representing better quality of life.
Change in Nociceptive Pain | 12 months post-completion of endotherapy
  Pain will be assessed using the PROMIS Nociceptive Pain Quality scales. Pain will be assessed before and after endotherapy (1, 3, 6, and 12 months). This pain scale goes from 5-25 with higher scores denoting worse pain.
Change in Neuropathic Pain | 12 months post-completion of endotherapy
  Pain will be assessed using the PROMIS Neuropathic Pain. Pain will be assessed before and after endotherapy (1, 3, 6, and 12 months). This pain scale goes from 5-25 with higher scores denoting worse pain.
Change in Pain Catastrophizing | 12 months post-completion of endotherapy
  Pain will be assessed using the UW Concerns about Pain Scale. Pain will be assessed before and after endotherapy (1, 3, 6, and 12 months). This pain scale ranges from 6 to 30 with higher scores denoting worse pain.
Change in Self-Efficacy | 12 months post-completion of endotherapy
  Pain will be assessed using the Self-Efficacy Scale Short Form. Pain will be assessed before and after endotherapy (1, 3, 6, and 12 months). This pain scale ranges from 6 to 30 with higher scores denoting worse pain.
Change in Chronic Pancreatitis-specific Pain | 12 months post-completion of endotherapy
  Pain will be assessed using the Comprehensive Pain Assessment Tool Short Form for Chronic Pancreatitis (COMPAT). Pain will be assessed before and after endotherapy (1, 3, 6, and 12 months). The COMPAT Short Form carries several sub-scores for pain pattern, pain severity, pain provocation, pain spreading, and pain description. The pain pattern scale ranges from 50-100 with higher scores denoting worse pain. The provocation score ranges from 0-70 with higher scores denoting worse pain. The severity score ranges from 0-100 with higher scores denoting worse pain. The spreading score ranges from 0-90 with higher scores denoting worse pain. The description score ranges from 0-80 with higher scores denoting worse pain. The total score ranges from 15-90 with higher scores denoting worse pain.
Quantitative Sensory Testing | The quantitative sensory testing will be assessed only once during the subject's baseline enrollment.
  Pancreatic Quantitative Sensory Testing (QST) will be assessed once during the baseline enrollment in the study. The QST provides Z-scores. The Z-scores range from 0 to -1.96 with 0 representing a normal score and -1.96 representing more widespread sensitization.
Pancreatic Endocrine Function via HbA1c | 12 months post-completion of endotherapy
  Pancreatic endocrine function will be assessed using the HbA1c. These will be measured before and after endotherapy (12 months). This is expressed as a % with higher values representing worse glycemic control.
Insulin Resistance | 12 months post-completion of endotherapy
  Pancreatic endocrine function will be assessed using a HOMA-IR score to assess the degree of insulin resistance. These will be measured before and after endotherapy (12 months). This score assesses insulin resistance by calculating the ratio between the serum insulin level and the fasting glucose level. Higher scores denote worse insulin resistance.
Insulin Sensitivity | 12 months post-completion of endotherapy
  Pancreatic endocrine function will be assessed using the QUICKI score, which measures the degree of insulin sensitivity. These will be measured before and after endotherapy (12 months). This is calculated using the ratio of fasting insulin and glucose. Lower levels denote worse insulin sensitivity.
Pancreatic Exocrine Function | 12 months post-completion of endotherapy
  Pancreatic exocrine function will be assessed using endoscopic pancreatic function testing. This will be performed before endotherapy and at 12 months post-endotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available to other researchers after completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available 24 months after study completion
Access Criteria: Investigators requesting data may request access to the data by contacting the study investigators.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT05012150/Prot_SAP_000.pdf